Diagnostic accuracy of a new ultrasound software compared to liver biopsy for Non Alcoholic Fatty Liver Disease (NAFLD) and Non Alcoholic Steato Hepatitis (NASH) in morbidly obese candidate to bariatric surgery and/or cholecystectomy.

Diagnostic accuracy of a new ultrasound software compared to liver biopsy for Non Alcoholic Fatty Liver Disease (NAFLD) and Non Alcoholic Steato Hepatitis (NASH) in morbidly obese candidate to bariatric surgery and/or cholecystectomy. Pilot study.

### PILOT PROSPECTIVE STUDY

#### 1. STUDY DIRECTOR

Prof. Gianfranco Silecchia, Direttore UOC Chirurgia Generale e Centro di Eccellenza in Chirurgia Bariatrica e Metabolica Sicob – Dipartimento di Scienze e biotecnologie medico-chirurgiche, "Sapienza" Università di Roma – Polo Pontino – gianfranco.silecchia@uniroma1.it;

### RESEARCHERS

- Dott.ssa Anna Guida, resident in General Surgery, University of Rome "La Sapienza" Polo Pontino
   Dipartimento di Scienze e biotecnologie medico-chirurgiche anna.guida@uniroma1-it
- 3. Dr. Piero Maceroni, CADI (Centro Alta diagnostica Immagini) director ICOT piero.maceroni@gmail.com
- 4. Prof. Vincenzo Petrozza, Direttore UOC Anatomia Patologica- Dipartimento di Scienze e biotecnologie medico-chirurgiche, "Sapienza" Università di Roma Polo Pontino vincenzo.petrozza@uniroma1.it
- 5. Prof.ssa Annarita Vestri, Dipartimento Sanita' Pubblica e malattie infettive, Sapienza-

"Sapienza" Università di Roma – Polo Pontino - annarita.vestri@uniroma1.it

The present has been financed within the framework of "Progetti per Avvio alla Ricerca – Tipo 2"

Year 2018, Sapienza University of Rome.

Research manager: Dr. Anna Guida,

Reference tutor: Professor Gianfranco Silecchia

## **Introduction**

The non-alcoholic fatty liver disease (NAFLD) is a systematic disease characterized by the presence of at least 5% of liver tissue, in the absence of other known causes of hepatopathy. To the present day, the NAFLD represents the first chronic hepatopathy cause. (1) It is a benign clinical condition that might evolve in non-alcoholic steato hepatitis (NASH) if inflammation and fibrosis occur along with the hepatic steatosis, with possible evolution in hepatic cirrhosis (in 25-30% of cases) and, subsequently, in hepatocellular carcinoma (7%) (2, 3).

The pathophysiological mechanisms that foster the progression from simple steatosis to NASH are complex and still not entirely clarified. It is certain that multiple genetic factors and acquired factors – such as insulin resistance, high ferritin and adiponectin reduction) are involved. NAFLD prevalence is directly proportional to obesity: it is estimated that 30% of the US population and 24% of the European population is affected by NAFLD and that within the obese population candidate to bariatric surgery the prevalence is at 90%. (4) In the western world, the prevalence of type 2 diabetes patients is at 60-70%. NAFLD shows a strong association with all the components of the metabolic syndrome, enough to be considered the hepatic manifestation of the metabolic syndrome (5).

Key elements of the NAFLD pathogenesis are hyperinsulinemia and insulin resistance. Insulin has three main actions in the liver: it increases glycogen synthesis, inhibits gluconeogenesis, and promotes lipogenesis. In patients with NAFLD, insulin resistance determines:

- 1) An increase in lipolysis in adipose tissue, resulting in increased circulating levels of free fatty acids, which convey to the liver level;
- 2) A reduction in glycogen synthesis and an increase in gluconeogenesis in the liver.

In response to insulin resistance, the body produces higher levels of insulin, which further increase liver lipogenesis, resulting in an intrahepatic accumulation of lipids and increased liver secretion of triglycerides in the form of VLDL lipoproteins.

In hepatocytes, the infestation of lipids causes a lipotoxicity that further worsens insulin resistance, increases oxidative stress and promotes inflammation and fibrosis (6,7).

The diagnosis of NAFLD is based on the combination of a number of clinical and radiological features. Hepatic enzymes are not a diagnostic criterion, as more than 60% of NAFLD patients and normal GPT values may have advanced degrees of steatohepatitis and 53% of NAFLD and increased GPT patients do not have NASH. Hepatic enzyme levels, therefore, are not reliably correlated with liver histology (8). Currently, validated methods for quantization of fibrosis, steatosis and hepatic necroinflammatory phenomena are: Elastography for the evaluation of hepatic fibrosis(9), contrastless MRI (10,11) or ecoguidated percutaneous biopsy for the evaluation of hepatic steatosis (12), ecoguidated percutaneous biopsy for the evaluation of necroinflammatory phenomena (13).

The NAFLD Activity Score (NAS) is the most widely used validated classifications for staging the NAFLS from a histological point of view(14), which assigns a score based on the following parameters:

- The steatosis level (with a score from 0 to 3)
- The degree of lobular inflammation (with a score from 0 to 3)
- The degree of balloning, i.e. hot air balloon hepatocytes (with a score from 0 to 2) According to the score, we can distinguish among:
- NAS 0 patients: with NAS Score < 3, in which the diagnosis of steatohepatitis is excluded (NO NASH)
- NAS 1 patients: with NAS Score between 3 and 4, indicative of probable pathology or borderline
- NAS 2 patients: with NAS Score ≥ 5 where steatohepatitis (NASH) diagnosis is made

# Purpose of the pilot study:

Evaluate the diagnostic accuracy of the new ultrasound software vs. liver histology, current reference standard for the diagnosis of NAFLD and NASH in obese patients (BMI > 30) candidates for bariatric laparoscopic surgery and/or cholecystectomy.

## **Type of study:**

Monocentric, open, sequential enrollment pilot study of 20 patients.

Datas will be analyzed with descriptive statistics, absolute values and percentages of concurrent and conflicting cases according to the two methods.

The concordance between the new ultrasound method and the liver biopsy will be evaluated and tested by the Monemar test

As the pilot study is used to assess whether there is good agreement between the two methods and in case of clinically significant response a study will be set up diagnostic with formal calculation of the sample size, with adequate power statistics and level of significance.

#### Inclusion criteria:

- 1. Patients who are candidates for bariatric surgery and are between 18 and 65 years of age,
- BMI > 40 kg/m2, in the absence of any other comorbidity
- BMI > 35 kg/m2, in the presence of comorbidities among those classically considered as associated with obesity (tab,) (15)

| Metabolic disease | Neoplasm | |
|---|---|---|
| Type 2 Diabetes Mellitus | Breast cancer | Esophageal cancer |
| Dyslipidemia | Pancreas cancer | Gallbladder cancer |
| Hyperuricemia and Gout | Colorectal cancer | Renal cancer |
| Female infertility | Prostate cancer | Leukemia |
| Polycystic ovary syndrome | Endometrial cancer | Ovarian cancer |
| | Liver cancer | |
| Cardiovascular Disease | Others | |
| Arterial Hypertension | Bronchial asthma | Psychological disorders |
| Coronary heart disease | Obstructive sleep apnea syndron | ne Gastroesophageal reflux |
| Congestive heart failure | Non alcoholic steatohepatitis | Urinary incontinence |
| Pulmonary embolism | Gallbladder disease | Osteoarthritis |
| Stroke | Intertrigo | Plantar fasciitis |

- ICM > 30 kg/m2, in the presence of T2DM not in glycomethabolic compensation
- 2. Patients who are candidates for laparoscopic cholecystectomy for symptomatic calculosis with BMI

#### **Exclusion criteria:**

- Age  $\leq 18$  or  $\geq 65$
- Any concomitant surgical procedure except cholecystectomy and repair of iatal hernia
- Conversion into laparotomic surgery
- Post-operative complications requiring new surgical treatment
- Non-compliant patient in follow-up

## **Methods:**

## **Pre- and post-operative evaluations:**

All patients will sign an informed consent ad hoc

Patients will be enrolled according to the PDTA deposited at the Health Directorate of the ICOT

Before surgical treatment all patients will be subjected to:

- standard liver ultrasound, shear wave elastography, attenuation imaging, shear wave dispersion blood tests: coagulation, GOT, GPT, GGT, alkaline phosphatase, total and fractionated bilirubin, fractionated cholesterol, triglycerides, insulinemia, glycaemia, Cpeptide

## **Imaging:**

The software is designed to be used on the Aplio i800 TUS system. (already supplied by our structure) and detects the attenuation that the signal ultrasound meets crossing the hepatic parenchyma and expresses this attenuation in Decibels on cm of hepatic parenchyma as a function of frequency (dB/cm/MHz) in a ROI of analysis.

Non-homogeneous zones are automatically excluded from the calculation. Being a newly introduced software, there is no reference standard with respect to the ultrasound systems currently used for the analysis of hepatic steatosis as the transient elastography (Fibroscan, Echosense Paris) or the CAP (Controlled AttenuationParameter).

There are no studies carried out with this software to date.

The methods that will be used are as follows:

## **Shear Wave Elastography (SWE)**

It quantifies the degree of liver fibrosis by measuring the speed of propagation of SW A focused ultrasonic pulse generates a tissue movement that creates shear waves (SW). The speed of movement of the shear waves depends on the rigidity of the crossed tissues.

Its tracking makes it possible to evaluate the rigidity of the tissue (the speed, expressed in m/s, is converted into "stiffness", expressed in kPa, using Young's equation).

# **Attenuation Imaging (AI)**

Quantifies the ultrasound attenuation of the tissue as an indicator of liver steatosis

Ultrasonic waves in the body are attenuated by sound loss, reflection and absorption (heat). Attenuation is frequency-dependent.

Attenuation Imaging is based on the RF information generated by the probe during conventional B-mode examination. The system compares the amplitude of the signal transmitted by the transducer with the return signal from the tissues at different depths, removing from the return ultrasound information all those pre- and post-processing compensations that the system introduces precisely to avoid having an uneven image between surface and depth. This analysis is carried out in a specific region of interest that the operator places on the tissue that is being analyzed. The value obtained represents the attenuation in Decibels per cm as a function of the transmission frequency used (dB/cm/MHz).

## **Shear Wave Dispersion (SWD)**

SWE has some limitations in the presence of steatosis and inflammation because it starts from the assumption that the liver is perfectly elastic.

Increasing the viscosity of the liver (inflammation, steatosis, circulation disorders) increases the phenomena of dispersion.

SWD measures the frequency dispersion of the shear wave propagation in the viscoelastic liver

The dispersion quantification ((m/s)/kHz) allows estimation of liver viscosity

SW signals are converted to SW frequencies with FFT (Fast Fourier Transform) processing

Increasing the viscosity (Pa\*s) with constant elasticity (kPa)-> the dispersion increases (steepest slope of the curve).

## Surgical technique:

All patients will undergo bariatric surgery according to the standard procedures validated by SICOB (15) and wedge resection of 1.5 cm x 1.5 cm at the level of the left hepatic lobe. In routine surgical practice, a liver biopsy is indicated in cases of hepatomegaly and clinical radiological suspicion of steatosis (16).

# Histology:

Histological examination of liver tissue will be performed on material from liver biopsy, fixed in formalin, included in paraffin and finally dissected. The reading of the set preparations will be performed by an expert pathologist who will not have access to the identity, clinical history and biochemical parameters of the patients.

A minimum biopsy sample length of  $1.5 \times 0.8$  cm. or at least 10 complete portal spaces will be required, it is strongly recommended whenever clinically possible to have a separate core for inclusion in cryomold and freezing at -80 C so as to have additional tissue available for possible molecular biology studies.

For liver histology sections of 3-4 µm will be obtained by staining with Hematoxylin/Eosin, PAS, PERLS, Gomoric Reticulum and Masonic Trichrome. NASH will be diagnosed according to Brunt's criteria (17). The NAFLD activity score (NAS) and a staging score capable of quantifying the extent of fibrosis in order to perform statistical correlations will be calculated (17). In addition, patients will be stratified according to the SAF score into no NAFLD, NAFLD or NASH (18).

### **References:**

- 1. Charlton MR, Burns JM, Pedersen RA, et al. Frequency and outcomes of liver transplantation for nonalcoholic steatohepatitis in the united states. Gastroenterology 2011;141:1249–53.
- 2. Rotonya M. Carr, Amanke Oranu, Vandana Khungar. Nonalcoholic Fatty Liver Disease. Pathophysiology and Management. Gastroenterology Clinic of North America 2016 Dec;45(4):639-652.)
- 3. Bugianesi E, Leone N, Vanni E *et al.* Expanding the natural history of nonalcoholic steatohepatitis: from cryptogenic cirrhosis to hepatocellular carcinoma. Gastroenterology 2002;123:134–40
- 4. Naga Chalasani, , Zobair Younossi, et al. The Diagnosis and Management of Non-alcoholic Fatty Liver Disease: Practice Guideline by the American Association for the Study of Liver Diseases, American College of Gastroenterology, and the American Gastroenterological Association. *Am J Gastroenterol* 2012; 107: 811–826; doi:10.1038/ajg.2012.128; published online 29 May 2012
- 5. Gao B, Tsukamoto H. Inflammation in alcoholic and nonalcoholic fatty liver disease: friend or foe? Gastroenterology 2016;150:1704–9.
- 6. Cosgrove D, Piscaglia F, Bamber J et al. EFSUMB guidelines and recommendations on the clinical use of ultrasound elastography. Part 2: Clinical applications. Ultraschall Med. 2013 Jun;34(3):238-53. doi: 10.1055/s-00331335375. Epub 2013 Apr 19).
- 7. Myers RP, Pomier-Layrargues G, Kirsch R et al. Feasibility and diagnostic performance of the FibroScan XL probe for liver stiffness measurement in overweight and obese patients. Hepatology. 2012 Jan;55(1):199-208. doi: 10.1002/hep.24624. Epub 2011 Nov 18)
- 8. Dyson JK, McPherson S, Anstee QM. Non-alcoholic fatty liver disease: non-invasive investigation and risk stratification. J Clin Pathol. 2013 Dec;66(12):1033-45. doi: 10.1136/jclinpath-2013-201620. Epub 2013 Aug 12).
- Lăpădat AM, Jianu IR et al. Non-invasive imaging techniques in assessing non-alcoholic fatty liver disease: a current status of available methods. Journal of Medicine and Life Vol. 10, Issue 1, January-March 2017
- Idilman IS, Aniktar H, Idilman R, Kabacam G, Savas B, Elhan A, Celik A, Bahar K, Karcaaltincaba M. Hepatic steatosis: quantification by proton density fat fraction with MR imaging versus liver biopsy. Radiology. 2013; 267:767-75.
- 11. Raptis DA, Fischer MA, Graf R, Nanz D, Weber A, Moritz W, Tian Y, Oberkofler CE, Clavien PA. MRI: the new reference standard in quantifying hepatic steatosis? Gut. 2012; 61:117-27
- 12. Angulo P. Nonalcoholic fatty liver disease. N Engl J Med 2002;346(16):1221–1231.

- 13. Angulo P, Keach JC, Batts KP, Lindor KD. Independent predictors of liver fibrosis in patients with nonalcoholic steatohepatitis. Hepatology 1999;30(6):1356–1362.
- 14. Pierre Bedossa, Keyur Patel Biopsy and Non-invasive Methods to Assess Progression of Nonalcoholic Fatty Liver Disease. Gastroenterology (2016), doi: 10.1053/j.gastro.2016.03.008.
- Diego Foschi, Maurizio De Luca, Giuliano Sarro, Paolo Bernante, Marco Antonio Zappa, Roberto Moroni, Giuseppe Navarra, Mirto Foletto, Valerio Ceriani, Luigi Piazza, Nicola Di Lorenzo LINEE GUIDA DI BUONA PRATICA CLINICA NELLA SELEZIONE, NELLA PREPARAZIONE, NEL TRATTAMENTO PERIOPERATORIO E A LUNGO TERMINE DEL PAZIENTE OBESO SOTTOPOSTO A CHIRURGIA BARIATRICA (2016)
- 16. Routine Liver Biopsy During Bariatric Surgery: an Analysis of Evidence Base. Mahawar KK, Parmar C, Graham Y, Abouleid A, Carr WR, Jennings N, Schroeder N, Small PK. Obes Surg. 2016 Jan;26(1):177-81
- 17. <u>Kleiner DE<sup>1</sup>, Brunt EM</u>. Nonalcoholic fatty liver disease: pathologic patterns and biopsy evaluation in clinical research. <u>Semin Liver Dis.</u> 2012 Feb;32(1):3-13. doi: 10.1055/s-0032-1306421. Epub 2012 Mar 13.
- 18. <u>Bedossa P<sup>1</sup>, Poitou C</u>. Histopathological algorithm and scoring system for evaluation of liver lesions in morbidly obese patients. Hepatology. 2012 Nov;56(5):1751-9. doi: 10.1002/hep.25889.